CLINICAL TRIAL: NCT03241212
Title: Adolescent Self-Care and Knowledge Education in Diabetes--Improved by Texting (ASKED-IT)
Brief Title: Adolescent Self-Care and Knowledge Education in Diabetes--Improved by Texting
Acronym: ASKED-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-1135
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: adolescent; young adult; knowledge; self-care
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): At baseline enrollment: participants will be asked to fill out a demographic survey, the MWIKAD survey and the SMOD-A survey. HbA1c, frequency of Blood Glucose (BG) checks and percent of glucose values above, within and below the target range will be extracted from chart review.
  Surveys (with the exception of demographics) and chart extraction will be repeated at 3 months and 6 months post enrollment.
- Texting (Experimental): Participants will be asked to complete the same surveys on the same timeline as above. The texting group will be asked to provide their cell phone number to the texting software.
  From baseline appointment to 26 weeks post enrollment, participants will receive a text message every Monday, Wednesday and Friday. Some text messages will be informational only, others will ask the participant for a response to a multiple-choice question with immediate feedback on the answer chosen.
  Interventions: Behavioral: Texting

INTERVENTIONS:
Behavioral: Texting — From baseline appointment to 6 month follow up, those participants randomly assigned to the texting intervention will receive a text message every Monday, Wednesday and Friday. Some text messages will be informational only, others will ask the participant for a response to a multiple-choice question with immediate feedback on the answer chosen.
  Arms: Texting

SUMMARY:
This study is a randomized controlled trial assessing diabetes knowledge (using a Mercy-What I Know About Diabetes Test (MWIKAD) validated survey) and self-care practices (using a validated Self-management of Type 1 Diabetes-Adolescence (SMOD-A) survey) at baseline, 3 months and 6 months. The intervention group will receive a minimum of 78 text messages related to diabetes over the course of 26 weeks from study enrollment. Subjects are invited to respond to some text messages which will be in the form of a multiple-choice question and if they do, they will receive an additional text message in response to their answer.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 1 diabetes mellitus
2. Receiving care in the pediatric clinic at the Barbara Davis Center (BDC)
3. Age 15-20 at study enrollment
4. English literate and English speaking
5. Ability to complete the required surveys
6. Have a personal cell phone with service compatible with EZTexting Platform
7. Able to provide informed assent or consent (if 18 years of age or older) and parental informed consent (if needed).

Exclusion Criteria:

1. Not planning to continue care in the pediatric clinic at BDC for at least the next 6 months.
2. Diabetes Diagnosis other than Type 1 Diabetes
3. Inability for the adolescent to respond to text messages (e.g. due to developmental delay)

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 148 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Change in knowledge about type 1 diabetes | 6 months from intervention
  Measured by the Mercy-What I Know About Diabetes Test (MWIKAD)

SECONDARY OUTCOMES:
Change in diabetes self-care practices | at 3 months and 6 months
  Assessed by the Self-Management of Type 1 Diabetes in Adolescents (SMOD-A) tool
Change in Hemoglobin A1c | at 3 months and 6 months
Change in blood glucose testing frequency | at 3 months and 6 months
Change in percent of blood glucoses high, in range and low | at 3 months and 6 months
Percent of text messages responded to in the study. | After 6 months of texting intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sonalee Ravi, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Barbara Davis Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No